CLINICAL TRIAL: NCT00283595
Title: Effect of Supraphysiological rhGH on Bone Metabolism in Patients With Anorexia Nervosa
Brief Title: Effect of Growth Hormone on Bone Metabolism in Anorexia Nervosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2005-P-001443/3; MGH
Record Dates: First submitted 2006-01-27; First posted 2006-01-30 (Estimated); Results first posted 2012-10-16 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Anorexia Nervosa; Osteopenia; Osteoporosis; Eating Disorders
Keywords: Anorexia Nervosa; Eating disorder; Bone; Growth hormone; Osteopenia; Osteoporosis
MeSH Terms: conditions — Anorexia Nervosa; Bone Diseases, Metabolic; Osteoporosis; Feeding and Eating Disorders | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Treatment with rHGH
  Interventions: Drug: Recombinant Human Growth Hormone
- 2 (Placebo Comparator): Treatment with Placebo
  Interventions: Drug: Placebo for Recombinant Human Growth Hormone

INTERVENTIONS:
Drug: Recombinant Human Growth Hormone — Dosage increased in steps for first four weeks. Self injection qd x 12 weeks
  Other Names: Nutropin AQ
  Arms: 1
Drug: Placebo for Recombinant Human Growth Hormone — Administered as Arm 1, rHGH active Injection qd x 12 weeks Dosage increase over four weeks
  Other Names: Placebo for Nutropin AQ
  Arms: 2

SUMMARY:
Decreased bone strength is a serious medical problem present in many women with Anorexia Nervosa, or disordered eating. Women with weaker bones are more likely to suffer broken bones than women with normal bone strength.

We are investigating whether a hormone that is naturally produced by the human body, called growth hormone, can help strengthen the bones of women with this type of disordered eating.

DETAILED DESCRIPTION:
* Twelve week study
* Eight visits, six of which can be conducted at your home physician's office
* Two bone density scans
* Hormonal and nutritional evaluations

ELIGIBILITY:
Inclusion Criteria:

* women between 14 to 45 years with anorexia nervosa

Exclusion Criteria:

* pregnancy
* previous history of malignancy.
* oral contraceptive pills or other hormones within last 8 - 12 weeks
* medications known to affect bone within last 12 weeks
* fracture within last 6 months

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Klibanski, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusettes General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were referred from by local eating disorders providers and were recruited from on-line advertisements. Recruitment period: April 2006 through November 2008.
Groups:
- Recombinant Human Growth Hormone(Subcutaneous Daily Injection): Treatment with rHGH
- Placebo (Subcutaneous Daily Injection): Treatment with Placebo
Period: Overall Study
Arm/Group | Recombinant Human Growth Hormone(Subcutaneous Daily Injection) | Placebo (Subcutaneous Daily Injection)
Started | 10 | 11
Completed | 9 | 9
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Recombinant Human Growth Hormone Group: Treatment with rHGH
- Placebo Group: Treatment with Placebo
- Total: Total of all reporting groups
Arm/Group | Recombinant Human Growth Hormone Group | Placebo Group | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (6.7) | 29.2 (8.6) | 28.7 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Bone Metabolism
Description: Change in the marker of bone formation, N-terminal pro peptide of type 1 procollagen (P1NP) levels, between baseline and 12 weeks
Time Frame: Baseline, 12 weeks
Population: Only subjects who completed study visits after the baseline visit were included in the analysis. The three subjects who discontinued the study only completed a baseline visit and were therefore not included in the analysis.
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Recombinant Human Growth Hormone Group | Placebo Group
Number analyzed (Participants) | 9 | 9
ng/ml | 34.3 (16.7) | 10.4 (7.1)

2. Secondary Outcome: IGF-1 Level
Description: Change in IGF-1 level between baseline and 12 weeks
Time Frame: Baseline, 12 Weeks
Population: The analysis group consisted of individuals who completed study visits after the baseline visit. The three subjects who did not continue in the study discontinued their participation after the baseline visit.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Recombinant Human Growth Hormone Group | Placebo Group
Number analyzed (Participants) | 9 | 9
ng/ml | 6.5 [-23.3 to 66.5] | 10 [-16.3 to 32]

ADVERSE EVENTS:
Arm/Group | Recombinant Human Growth Hormone Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 8/10 | 9/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Human Growth Hormone Group (N=10) | Placebo Group (N=11)
Constipation (Gastrointestinal disorders) | 3 (4) | 5 (12)
Arthralgias (Musculoskeletal and connective tissue disorders) | 2 (4) | 2 (3)
Headache (Nervous system disorders) | 5 (9) | 4 (5)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 4 (7)
Edema (General disorders) | 4 (4) | 1 (2)
Lightheadedness (General disorders) | 3 (6) | 5 (7)
Polyuria (Endocrine disorders) | 2 (2) | 0 (0)
Depressive symptoms (Psychiatric disorders) | 2 (2) | 4 (6)
Nausea (Gastrointestinal disorders) | 3 (6) | 3 (3)
Irritation at injection site (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (4)
Blurry vision (Eye disorders) | 1 (1) | 0 (0)
Paresthesias (carpal tunnel symptoms) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (3)
Cold intolerance (General disorders) | 0 (0) | 3 (6)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Polydypsia (General disorders) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No